CLINICAL TRIAL: NCT03797092
Title: Stem Cell Therapy in Non-IschEmic Non-treatable Dilated CardiomyopathiEs II: a Pilot Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JKastrup (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor-Investigator, JKastrup, Professor, Doctor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCIENCE II - Pilot
Record Dates: First submitted 2018-06-28; First posted 2019-01-08 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Non-ischemic Dilated Cardiomyopathy
Keywords: Stem cell therapy; Heart failure; Clinical trial; Allogeneic
MeSH Terms: conditions — Heart Failure | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Open randomized treatment group and control group clinical trial
Who Masked: Outcomes Assessor
Masking Description: The patients will be randomized to either IMP or control in a 2:1 randomization.
  The outcome ECHO investigations will be analyzed blinded by an independent core lab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Allogeneic adipose-derived stromal cells (CSCC_ASC)
  Interventions: Biological: Allogeneic adipose-derived stromal cells (CSCC_ASC); Other: Control group
- Control group (No Intervention): No treatment

INTERVENTIONS:
Biological: Allogeneic adipose-derived stromal cells (CSCC_ASC) — Active group
  Other Names: Investigational medicinal product
  Arms: Active
Other: Control group — No treatment
  Arms: Active

SUMMARY:
The overall aim of the project is to test the feasibility and safety of allogeneic adipose-derived stromal cells (CSCC_ASC) investigational medicinal product, to improve myocardial function in patients with non-ischemic dilated cardiomyopathies (NIDCM) and heart failure.

DETAILED DESCRIPTION:
Study design

The primary objective of the study is to investigate safety and regenerative capacity of direct intra-myocardial injection of 100 million allogeneic CSCC_ASCs in NIDCM patients with reduced left ventricular EF (≤ 40%) and heart failure.

It is a proof of concept study enrolling a total of 30 NIDCM patients with heart failure who will be randomly allocated in a 2:1 ratio to either CSCC_ASC cell therapy (Stem Cell Group) or no cell therapy (Control Group). The treatment period is estimated to be 6 months (efficacy end-point) with a 12-month follow-up period for safety end-points.

Patient treatment and follow-up

* The cell IMP will be delivered by a courier service to from REGIONH to UKCL using validated portable dry liquid nitrogen shipping containers. It will then be stored in nitrogen vapour containers until treatment.
* The preparation of the IMP will be performed as described in the treatment manual. The IMP will be thawed and prepared for injection immediately before treatment.
* A 3-D map of the left ventricle will be created using the NOGA XP® system (Biological Delivery System, Cordis, Johnson & Johnson, USA). The delivery of the IMP (100 million ASCs) into the myocardium will be performed by 10-15 injections of 0.2 cc, as described in the treatment manual.
* The post cell therapy surveillance will include clinical and laboratory safety follow-up with monitoring of cardiac enzymes, hemodynamic and rhythm stability. The clinical follow-up will be obtained at pre-defined time points. The presence of allogeneic HLA anti-bodies will be monitored three and six months after treatment. End-points will be monitored continuously and reported as occurring throughout the 12 months follow-up period.

Primary and secondary endpoints

The primary endpoint is change in left ventricle end-systolic volume (LVESV) at 6 months follow-up measured by Echocardiography.

The secondary endpoints are safety evaluated by development of allogeneic antibodies and laboratory safety measurements 1, 3 and 6 months after treatment and changes in left ventricular ejection fraction (LVEF), end-diastolic volume and myocardial mass at 6 months follow-up.

Additional secondary endpoints are changes in NYHA, Kansas City Cardiomyopathy Questionnaire, EQ-5D3L Questionnaire, 6 min walking test, additional echocardiographic measures (Global strain %) and NT-pro-BNP.

Safety of allogeneic CSCC_ASCs with respect to incidence and severity of serious adverse events and suspected unrelated serious adverse events will be evaluated at 12 months follow-up.

Outcome measures for safety Safety endpoints will be collected, reported to the authorities and monitored according to legislation during the entire study period.

Adverse event (AE) is defined as any untoward medical occurrence in a subject who was treated with an investigational product, and does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease, whether or not related to the investigational product.

Serious adverse event (SAE) is defined as any untoward medical occurrence that:

1. results in death
2. is life-threatening
3. requires inpatient hospitalisation or prolongation of existing hospitalisation
4. results in persistent or significant disability/incapacity
5. is a congenital anomaly/birth defect
6. is medically important

Suspected unexpected serious adverse event reactions (SUSAR) is defined as a SAE occurring in a subject in an interventional study that is assessed as both causally related to the suspect product under clinical investigation and unexpected per the Investigator's Brochure (IB).

An independent Data Safety Monitoring Board (DSMB) will be established to evaluate the safety of the treatment. The DSMB will report directly to the director of the Project Management Board, which will take the necessary action upon the DSMB's recommendations.

Study medication The investigational cell product, CSCC_ASC, will be produced in an approved GMP facility in Cardiology Stem Cell Centre at Rigshospitalet University Hospital, Copenhagen, Denmark.

The production of the allogeneic CSCC_ASCs will follow the description in an approved Investigational Medicinal Product Dossier. The cell product will come from healthy donors.

The production unit will label the investigational medicinal product (IMP) in accordance with the legislation and keep the randomisation code until finalisation of the clinical trial. The final cell products will be stored in nitrogen vapour containers until clinical use.

Allogeneic MSCs and ASCs have been administered to more than 600 patients with heart disease. In the conducted clinical trials there has not been any serious adverse event due to the treatment. A few patients have developed transient donor specific HLA-antibodies in serum within the first months after treatment. However, none of the patients had any symptoms related to the presence of antibodies. Transient fever was registered in a few patients, but it could as well be due to the treatment procedure or the disease for treatment.

Based on the accumulated safety and efficacy evidence with clinical use of allogeneic MSCs and ASCs in conducted clinical trials and the safety data from the CSCC_ASC phase I trial and the two ongoing phase II trials then it is concluded that it is safe to conduct a pilot CSCC_ASC trial in patients with NIDCM and HF.

Echocardiography

The echocardiography data will be recorded at pre-defined intervals according to American Society of Echocardiography (ASE) and European Association of Cardiovascular Imaging (EACVI) recommendations. For each patient at least five end-expiratory full cardiac cycles will be recorded for each protocol specified view. All acquired images will be de-identified and transferred to independent imaging core-lab (Stanford Cardiovascular Institute Clinical Biomarker & Phenotyping Core Lab). The recordings will be analyzed at the end of the study by an independent echocardiographer who will be blinded to the patient's treatment status and the timing of the recordings. All measurements will be performed according to ASE/EACVI recommendations. All echocardiographic measurements will be averaged over 5 cardiac cycles. Left ventricular end-systolic dimension (LVESD) and end-diastolic dimension (LVEDD) will be measured in the parasternal long-axis view. Left ventricular end-systolic volume (LVESV), left ventricular end-diastolic volume (LVEDV), and LVEF will be estimated using the Simpson's biplane method. Peak longitudinal strains will be computed automatically to generate regional data from each of the 17 segments and then averaged to calculate global longitudinal strain.

ELIGIBILITY:
Inclusion Criteria:

1. 30 to 80 years of age
2. Signed informed consent
3. Patients with non-ischemic dilated cardiomyopathy
4. NYHA ≥ II in spite of optimal heart failure treatment and have no other treatment options
5. Heart failure medication unchanged two months prior to inclusion/signature of informed consent. Changes in diuretics accepted
6. LVEF ≤ 405%
7. Plasma NT-pro-BNP > 300 pg/ml (> 35 pmol/L)
8. Patients cannot be included until three months after implantation of a cardiac resynchronisation therapy device (CRTD) and until 1 month after an ICD unit

Exclusion Criteria:

1. Heart Failure NYHA I
2. Moderate to severe aortic stenosis (valve area < 1.3 cm2) or valvular disease with option for surgery or interventional therapy.
3. Heart failure caused by cardiac valve disease or untreated hypertension.
4. If the patient is expected to be candidate for MitraClip therapy of mitral regurgitation in the 12 months follow-up period.
5. Cardiomyopathy with a reversible cause that has not been treated e.g. thyroid disease, alcohol abuse, hypophosphataemia, hypocalcaemia, cocaine abuse, selenium toxicity & chronic uncontrolled tachycardia
6. Cardiomyopathy in association with a neuromuscular disorder e.g. Duchenne's progressive muscular dystrophy
7. Previous cardiac surgery
8. Diminished functional capacity for other reasons such as: obstructive pulmonary disease (COPD) with forced expiratory volume (FEV) <1 L/min, moderate to severe claudication or morbid obesity
9. Clinical significant anaemia (haemoglobin < 6 mmol/L), leukopenia (leucocytes < 2 109/L), leucocytosis (leucocytes > 14 109/L) or thrombocytopenia (thrombocytes < 50 109/L)
10. Reduced kidney function (eGFR < 30 ml/min)
11. Left ventricular thrombus
12. Anticoagulation treatment that cannot be paused during cell injections.
13. Patients with reduced immune response
14. History with malignant disease within five years of inclusion or suspected malignity - except treated skin cancer other than melanoma
15. Pregnant women
16. Woman of childbearing potential unless βHCG negative and they should be on contraception during the trial
17. Other experimental treatment within four weeks of baseline tests
18. Participation in another intervention trial
19. Life expectancy less than one year

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricle end-systolic volume | 6 months after treatment
  Measured using echocardiography

SECONDARY OUTCOMES:
Allogeneic antibodies | Up to 12 months after treatment
  Development of allogeneic antibodies and laboratory safety measurements 1, 3 and 6 months after treatment
Left ventricular ejection fraction | 6 months after treatment
  Changes in LVEF
Myocardial mass of left ventricle | 6 months after treatment
  Change in echo measured global myocardial mass
NYHA | 6 months after treatment
  Symptoms
Kansas City Cardiomyopathy Questionnaire | 6 months after treatment
  Questionnaire
EQ-5D3L Questionnaire | 6 months after treatment
  Questionnaire
6 min walking test | 6 months
  Test

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Vrtovec, MD, PhD, Principal Investigator — Dep. of Cardiology, Uni. Medical Center Ljubljana, Slovenia
Locations (1):
- The Heart Centre, Rigshospitalet University Hospital Copenhagen,, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The entire study will be published and shared with other researchers

REFERENCES:
- [Result] Kastrup J, Haack-Sorensen M, Juhl M, Harary Sondergaard R, Follin B, Drozd Lund L, Monsted Johansen E, Ali Qayyum A, Bruun Mathiasen A, Jorgensen E, Helqvist S, Jorgen Elberg J, Bruunsgaard H, Ekblond A. Cryopreserved Off-the-Shelf Allogeneic Adipose-Derived Stromal Cells for Therapy in Patients with Ischemic Heart Disease and Heart Failure-A Safety Study. Stem Cells Transl Med. 2017 Nov;6(11):1963-1971. doi: 10.1002/sctm.17-0040. Epub 2017 Sep 7. PMID 28880460
- See also: PubMed abstract related to the used allogeneic stem cell product — https://www.ncbi.nlm.nih.gov/pubmed/28880460